CLINICAL TRIAL: NCT06698445
Title: Effect of Short Film Video Training Prepared for Children Undergoing Bone Marrow Aspiration and Biopsy on Children's Anxiety, Fear, Pain and Satisfaction
Brief Title: Effect of Short Film Video Training Prepared for Children Undergoing Bone Marrow Aspiration and Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-112
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anxiety and Fear; Pain; Satisfaction
Keywords: anxiety; fear; pain; satisfaction; children
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Patients who meet the sample selection criteria will be randomly and equally distributed into 2 groups (1st experimental group, 2nd control group) using a computer program according to gender, age and whether or not KIA has been applied for the first time, thus providing simple stratified randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Film Video (Experimental): The short film training video will be prepared by researchers based on literature and appropriate for the level of children aged 7-12. The content will include topics such as preparation for KİAB, KİAB environment and the process after KİAB. Since the short film will be shot in a realistic manner, the scenario will include a doctor, a nurse, a child patient and a parent. The short film will be shot in the clinic where the data will be collected, at the appropriate time for the clinic. After the short film is shot, the editing process will be done and the final version will be given.
  Interventions: Other: Short film video
- Control (No Intervention): The control group will be given verbal information as a routine clinical practice.

INTERVENTIONS:
Other: Short film video — The short film training video will be prepared by researchers based on literature and appropriate for the level of children aged 7-12. The content will include topics such as preparation for KİAB, KİAB environment and the process after KİAB. Since the short film will be shot in a realistic manner, the scenario will include a doctor, a nurse, a child patient and a parent. The short film will be shot in the clinic where the data will be collected, at the appropriate time for the clinic. After the short film is shot, the editing process will be done and the final version will be given.
  Arms: Short Film Video

SUMMARY:
In this study, it is aimed to examine the effect of short film video education given to children aged 7-12 years who will undergo CIAB before the procedure on the anxiety, fear, pain and satisfaction levels of the children. It will be carried out in a single-center, randomized controlled experimental design. The universe of the study will be children aged 7-12 who applied to the Children's Department of Mersin University Oncology and Hematology Hospital, and the sample will consist of 60 children who meet the criteria for inclusion in the study. In the collection of research data; Introductory Information Form, Child Anxiety Scale, Child Fear Scale, Numerical Pain Scale, Vital Signs Follow-up Form and Child Satisfaction Scale will be used.

DETAILED DESCRIPTION:
This study aims to examine the effects of short film video training given to children aged 7-12 years who will undergo CIAB before the procedure on the anxiety, fear, pain and satisfaction levels of the children. It will be carried out in a single-center, randomized controlled experimental design. The universe of the study will be children aged 7-12 who applied to the Children's Department of Mersin University Oncology and Hematology Hospital, and the sample will consist of 60 children who meet the criteria for inclusion in the study.

Introductory Information Form, Child Anxiety Scale, Child Fear Scale, Numerical Pain Scale, Vital Sign Follow-up Form and Child Satisfaction Scale will be used in the collection of research data.

Data Collection

* Data will be collected in the waiting room after the child is examined in the clinic. In the collection of data, the child patients and their parents who meet the inclusion criteria of the study and agree to participate in the study, will be informed about the purpose of the study and the research, and their verbal and written permissions will be obtained.
* Patients who meet the sample selection criteria will be randomly and equally distributed into 2 groups (1st experimental group, 2nd control group) via a computer program (http://www1.assumption.edu/users/avadum/applets/RandAssign/GroupGen.html).
* The data collection forms in the study (Introductory Information Form, Child Anxiety Scale, Child Fear Scale and Vital Signs Follow-up Form) will be applied to the children and parents in the sample group. The anxiety and fear assessment of the children will be carried out by the child, nurse and parent.
* A short film video training will be introduced to the children and parents in the experimental group and the children will be allowed to watch it on a tablet. After watching the short film video training, the children will be applied the CIAB procedure.
* The routine application of the clinic (verbal information) will be applied to the children and parents in the control group.
* After the CIAB procedure, the Child Anxiety Scale, Child Fear Scale, Numerical Pain Scale, Vital Signs Follow-up Form and Child Satisfaction Scale will be applied to all groups in the experimental and control groups. The anxiety, fear and pain assessment of the children will be carried out by the child, nurse and parent.

Statistical package program (SPSS 20) will be used in the analysis of the research data. The statistical significance level was determined as 0.05. The conformity of the data used to the normal distribution will be checked with kurtosis and skewness values. In the comparison of quantitative data with normal distribution, independent t test will be applied for the difference between two independent groups, and in the comparison of more than two dependent groups, variance analysis in repeated measurements will be applied, and in the case of a difference, Bonferroni will be used to find the group that made the difference. In the comparison of quantitative data with non-normal distribution, Mann Whitney U test will be applied for the difference between two independent groups, and in the comparison of more than two dependent groups, Friedman test will be applied, and in the case of a difference, corrected Bonferroni will be used to find the group that made the difference. Chi-square analysis will be applied to test the relationship between categorical variables. Cohen's Kappa Test will be applied in the inter-observer agreement analysis. In addition, at the end of the research, the status of working with a sufficient sample size will be tested with post-hoc power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 7-12
* The child will undergo bone marrow aspiration and biopsy
* The child will undergo bone marrow aspiration and biopsy for the first time
* Volunteering to participate in the study

Exclusion Criteria:

* Not being between the ages of 7-12
* Having another chronic disease
* Having a family member undergo bone marrow aspiration and biopsy
* Having a communication, mental or neurological problem

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Anxiety level | 1 hour
  Child Anxiety Scale: E This scale is for children ages 4-10. Children are told, "Imagine all your anxious or nervous feelings being in the bulb or bottom part of the thermometer" or "If you are a little anxious or tense, feelings may go up a little bit on the thermometer. If you are very, very anxious or tense, feelings may go all the way to the top. Put a line on the thermometer to show how anxious or nervous you are." To measure state anxiety, the child is asked to mark what he or she is feeling "right now."
Fear level | 1 hour
  Child Fear Scale: This scale includes 5 different facial expressions. This scale is scored between 0-4 and is stated to be a reliable and valid measurement tool in the assessment of fear.
Pain level | 1 hour
  Numerical Pain Scale, this method for determining the intensity of pain aims to have the patient describe his pain with numbers. In numerical scales, the absence of pain (0) is evaluated as unbearable pain (10).
Satisfaction level | 1 hour
  The Child Satisfaction Scale was developed by researchers in line with the literature in a way that child patients can easily understand. The numbers between 0 and 10, which children will indicate by circling the point corresponding to their satisfaction with the education provided, are placed on a horizontal line. A score of 0 on the scale indicates "not satisfied at all" and a score of 10 indicates "extremely satisfied". In addition, there is a visual reflecting the degree of satisfaction in the places where the points are located.

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Karakul, Principal Investigator — Tarsus University
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdolkarimi B, Zareifar S, Golestani Eraghi M, Saleh F. Comparison Effect of Intravenous Ketamine with Pethidine for Analgesia and Sedation during Bone Marrow Procedures in Oncologic Children: A Randomized, Double-Blinded, Crossover Trial. Int J Hematol Oncol Stem Cell Res. 2016 Oct 1;10(4):206-211. PMID 27928474
- [Background] Alonso Puig M, Alonso-Prieto M, Miro J, Torres-Luna R, Plaza Lopez de Sabando D, Reinoso-Barbero F. The Association Between Pain Relief Using Video Games and an Increase in Vagal Tone in Children With Cancer: Analytic Observational Study With a Quasi-Experimental Pre/Posttest Methodology. J Med Internet Res. 2020 Mar 30;22(3):e16013. doi: 10.2196/16013. PMID 32224482
- [Background] Baghele A, Dave N, Dias R, Shah H. Effect of preoperative education on anxiety in children undergoing day-care surgery. Indian J Anaesth. 2019 Jul;63(7):565-570. doi: 10.4103/ija.IJA_37_19. PMID 31391620
- [Background] Balasubramanian M, Sangoi NN. Utility of Bone Marrow Examination in Pediatric Age Group: Experience of a Tertiary Healthcare Centre in India. Cureus. 2022 Jul 20;14(7):e27056. doi: 10.7759/cureus.27056. eCollection 2022 Jul. PMID 36000100
- [Background] Bozkul G, Karakul A, Duzkaya DS, Dilsen S. Effect of short film video and video-based education on fear, pain, and satisfaction of children undergoing day surgery. J Pediatr Nurs. 2024 Mar-Apr;75:49-56. doi: 10.1016/j.pedn.2023.11.029. Epub 2023 Dec 14. PMID 38101311
- [Background] Bernier Carney KM, Jung SH, Iacob E, Lewis M, Linder LA. Communication of pain by school-age children with cancer using a game-based symptom assessment app: A secondary analysis. Eur J Oncol Nurs. 2021 Jun;52:101949. doi: 10.1016/j.ejon.2021.101949. Epub 2021 Mar 20. PMID 33813185
- [Background] Comparcini D, Simonetti V, Galli F, Saltarella I, Altamura C, Tomietto M, Desaphy JF, Cicolini G. Immersive and Non-Immersive Virtual Reality for Pain and Anxiety Management in Pediatric Patients with Hematological or Solid Cancer: A Systematic Review. Cancers (Basel). 2023 Feb 3;15(3):985. doi: 10.3390/cancers15030985. PMID 36765945
- [Background] Hoag JA, Karst J, Bingen K, Palou-Torres A, Yan K. Distracting Through Procedural Pain and Distress Using Virtual Reality and Guided Imagery in Pediatric, Adolescent, and Young Adult Patients: Randomized Controlled Trial. J Med Internet Res. 2022 Apr 18;24(4):e30260. doi: 10.2196/30260. PMID 35436209